CLINICAL TRIAL: NCT05145179
Title: A Phase I, Multicenter, Open-Label, First-in-Human Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Potential Anti-tumor Effects of SSGJ-705 in Patients With Advanced or Metastatic HER2-expressing Solid Tumors
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Potential Anti-tumor Effects of SSGJ-705 in Patients With Advanced or Metastatic HER2-expressing Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-705-ST-I-01
Record Dates: First submitted 2021-11-25; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-07

CONDITIONS: Receptor, ErbB-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HER2-expressing Solid Tumors (Experimental): SSGJ-705 Administered via intravenous (IV) infusion
  Interventions: Drug: SSGJ-705

INTERVENTIONS:
Drug: SSGJ-705 — 0.1, 1, 3, 6, 10, 15 or 20mg/kg, IV, Day 1, 8, 15 of each treatment cycle, up to disease progression or intolerable toxicity, death, early withdrawal from the study or loss to follow-up, withdrawal of consent, or the end of the treatment period, whichever occurs first. Every 4 weeks a treatment cycle.

SUMMARY:
The study will consist of two parts: a dose-escalation part (Part 1) and a dose expansion part (Part 2). In both study parts, SSGJ-705 will be administered，the administration duration may be adjusted based on outcomes of previous patients if necessary) followed by safety, PK, PD, potential anti tumor effects and immunogenicity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 year, male or female.
* Life expectancy ≥12 weeks (according to Investigator's judgement).
* Patients with histologically or cytologically confirmed locally advanced or metastatic non resectable HER2-expressing Solid Tumors
* Patients who have at least one measurable lesion (radiation-naïve) according to RECIST v1.1
* ECOG performance status 0-1
* Adequate organ and bone marrow function evaluated by laboratory tests
* Male patients who are surgically sterilized or who agree to use highly effective contraceptive measures during the study and for at least 6 months after administration of the last study drug dose
* Willing to provide written informed consent and willing and able to comply with all study procedures.

Exclusion Criteria:

* Receive chemotherapy, targeted therapy, or other antitumor therapy within 3 weeks prior to initial dosing
* Patients whose toxicity due to previous anticancer therapy has not been reduced to NCI CTCAE Grade 1 or lower, or any greater than NCI CTCAE 1 AE exists within 2 weeks before enrollment, not including hair loss and fatigue
* Patients requiring systemic systemic therapy with systemic hormones or other immunosuppressive agents within 4 weeks prior to initial administration and during the study period
* Previous cumulative doses of adriamycin > 720 mg/m2, adriamycin >360 mg/m2 or other cumulative doses of adriamycin were converted to equal doses of adriamycin >360 mg/m2
* Patients who underwent major surgery within 4 weeks of initial dosing and have not fully recovered or who plan to undergo major surgery during the trial
* In addition to palliative radiotherapy, other anticancer treatments not specified in the protocol are planned for the duration of the trial
* Always received total pelvic radiotherapy
* Had an active or prior autoimmune or inflammatory disease within the last 3 years prior to study treatment
* Severe disease of cardiovascular and cerebrovascular diseases
* History of active tuberculosis
* A history of (non-infectious) pneumonia/interstitial pneumonia or a history of present pneumonia/interstitial pneumonia requiring steroid treatment
* Severe dyspnea or the need for supplemental oxygen therapy at rest due to complications of advanced malignancy; Newly diagnosed or symptomatic central nervous system (CNS) metastasis, spinal cord compression, or cancerous meningitis
* Persons with a history of primary immunodeficiency disease, including but not limited to HIV-positive serum
* Hepatitis B virus (HBV) and hepatitis C virus (HCV) positive subjects
* Women/men who are pregnant or breast-feeding or planning to give birth
* A history of mental or substance abuse that may affect study compliance
* Allergy to other antibody drugs or to any excipients in the study drug
* Who received live vaccine within 30 days prior to initial administration (within 72 hours for COVID-19 vaccine), or who plan to receive any live vaccine during the study
* Previous organ and allogeneic stem cell transplants (except transplants that do not require immunosuppressive therapy, such as corneal and hair transplants)
* Participated in any medical device or drug clinical study within 1 month prior to screening
* The inestigators considered that this would significantly increase the risk of administration of the investigational drug, or that it would affect efficacy evaluation or other conditions requiring exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
DLT | At the end of Cycle 1 (each cycle is 28 days)
  Dose-limiting toxicity（part 1）
MTD | up to 1 years
  maximum tolerated dose（part 1）
RP2D | up to 1 years
  Objective response rate (ORR) per RECIST 1.1 criteria according to investigators recommended Phase II dose（part 1）
ORR | up to 1 years
  Objective response rate (ORR) per RECIST 1.1 criteria according to investigators assessment（part 2）

SECONDARY OUTCOMES:
Adverse events | up to 1 years
  the safety of SSGJ-705 in patients with advanced or metastatic HER2-expressing solid tumors who have failed standard treatment
Maximum Plasma Concentration (Cmax) | up to 1 years
  To evaluate the Cmax of single and multiple doses of SSGJ-705 in patients with advanced or metastatic HER2 expressing solid tumors who have failed standard treatments
Area Under the Curve (AUC) | up to 1 years
  To evaluate the AUC of single and multiple doses of SSGJ-705 in patients with advanced or metastatic HER2 expressing solid tumors who have failed standard treatments
incidence of anti-609A antibodies | up to 1 years
  incidence of anti-609A antibodies
Median Progression-free Survival (PFS) | up to 1 years
  The Kaplan-Meier method will be used to estimate median PFS.
Overall Survival (OS) | up to 1 years
  The Kaplan-Meier method will be used to estimate median OS.

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, PhD, Principal Investigator — The Fifth Medical Center of the People's Liberation Army; Ying Cheng, PhD, Principal Investigator — Jilin Provincial Cancer Hospital

IPD SHARING:
Plan to Share IPD: No